CLINICAL TRIAL: NCT01829503
Title: Phase II Study of Decitabine and Cytarabine for Older Patients With Newly Diagnosed AML
Brief Title: Phase II Study of Decitabine and Cytarabine for Older Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annie Im, M.D. (Other)
Responsible Party: Sponsor-Investigator, Annie Im, M.D., MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-099
Record Dates: First submitted 2013-03-06; First posted 2013-04-11 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Phase II; decitabine; cytarabine; older patients; newly diagnosed; AML; Newly Diagnosed AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Cytarabine; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- decitabine and cytarabine (Experimental)
  Interventions: Drug: decitabine and cytarabine; Other: Supportive Care

INTERVENTIONS:
Drug: decitabine and cytarabine
Other: Supportive Care — blood product transfusions, antiemetic medications, antiviral and antifungal medications, empiric antibiotics

SUMMARY:
Primary objective: To determine the efficacy of an induction regimen using decitabine as an epigenetic primer followed by cytarabine in the treatment of older patients with newly diagnosed Acute myeloid leukemia (AML).

Primary endpoint:

Complete remission rates

Secondary objective: To determine the safety of an induction regimen of decitabine followed by cytarabine in the treatment of older patients with newly diagnosed AML, evaluate survival and identify potential predictive factors for response to treatment

Secondary endpoints:

* Treatment related toxicities
* 4 and 8 week mortality
* Overall survival
* Relapse-free survival
* Predictive factors for response to treatment
* Quality of Life measures including self reported symptoms and assessment of sleep patterns

Treatment administration

Induction therapy Eligible patients will be treated with induction therapy (decitabine + cytarabine) at the University of Pittsburgh Cancer Center inpatient leukemia service at Shadyside Hospital. Patients will receive decitabine 20mg/m2 in 100mL normal saline (NS) intravenously (IV) over 1 hour daily for five days, followed by cytarabine 100mg/m2 in 1000 mL normal saline (NS) as a continuous IV infusion over 24 hours for 5 days. Treatment should be discontinued or delayed for any of the following during the treatment period: a rise in serum creatinine > 2x patient baseline or upper limit of normal (whichever is higher) unless there is an identifiable reversible etiology, or ALT, AST or total bilirubin > 5x upper limit of normal, and should be held until resolution below these parameters. There are no parameters for dose reduction.

Patients who have persistent disease on post-treatment bone marrow aspirate and biopsy, will undergo a repeat cycle of induction with decitabine followed by cytarabine as outlined above.

Supportive care including blood product transfusions, antiemetic medications antiviral and antifungal medications, or empiric antibiotics may be used at the clinical discretion of the provider.

Maintenance therapy Patients in complete response (CR) will proceed to decitabine maintenance therapy, where each treatment will be decitabine 20mg/m2 in 100mL normal saline (NS) intravenously (IV) over 1 hour daily for five days administered in the outpatient setting. Maintenance treatments will be continued until disease relapse. Maintenance treatments can be administered as an outpatient at the Hillman Cancer Center, or at a University of Pittsburgh Medical Center (UPMC) facility that is able to administer chemotherapy under the supervision of an Oncologist

Evaluations during maintenance Phase:

During maintenance therapy, complete blood count (CBC) w/ diff/platelets, CMP (Na, K, Cl, carbon dioxide (CO2), glucose, blood urea nitrogen (BUN), Cr, Ca, Total Protein, Albumin, AST, ALT, Alk Phos, Total Bilirubin) will be checked each cycle on day 14 [+/- 4 days].

Within 7 days of start of new cycle, study visits will include physical exam, adverse events assessment, CBC and comprehensive metabolic panel (CMP).

Maintenance cycles will be 28 days [+/- 7 days]. Cycles can be held up to 4 weeks [28 days]. For start of new cycle, any grade 3 or 4 non-hematologic toxicity possibly, probably or definitely related to decitabine therapy must resolve to grade 2 or baseline.

In addition the following lab parameters must be met to start a new cycle of maintenance:

Absolute Neutrophil Count (ANC) > or = 1000/mm3 Platelets >/= 50,000/mm3 AST or ALT < 2 x Uppler Limit of Normal (ULN) Total billirubin < 2 x ULN Serum creatinine < 2x patient baseline or upper limit of normal (whichever is higher)

[If lab parameters are not met for start of cycle, these labs will be checked a minimum of once per week]. If start of new cycle is held for more than 4 weeks [28 days], the subject will be off treatment.

Other reasons for delay in treatment should be discussed with the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70, or age ≥ 60 ineligible for treatment with standard induction chemotherapy (based on physician discretion or patient refusal), with a new diagnosis of AML based on World Health Organization Classification.
2. Eastern Cooperative Oncology Group Performance Status of 0-2
3. Cardiac ejection fraction ≥45%
4. Males are eligible to enter and participate in the study if they have either had a prior vasectomy or agree to avoid sexual activity or use adequate contraception from screening through two months post the last dose of decitabine

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia
2. Life expectancy ≤3 months
3. Prior use of any hypomethylating agent or cytarabine
4. Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy
5. Serum creatinine > 2x upper limit of normal
6. Aspartate aminotransferase (AST),alanine aminotransferase (ALT), or total bilirubin > 5x upper limit of normal
7. History of psychiatric disorder which may compromise compliance with the protocol or which does not allow for appropriate informed consent
8. Patient may not be receiving any other antineoplastic agents (hydroxyurea is allowed)
9. Concurrent malignancy. Exception: Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible. Subjects with second malignancies that are indolent or definitively treated may be enrolled.
10. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Im, MD, Principal Investigator — UPCI
Locations (1):
- University of PIttsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Im A, Quann K, Agha M, Raptis A, Redner RL, Hou JZ, Farah R, Dorritie KA, Sehgal AR, Normolle D, Bovbjerg DH, Aggarwal N, Herman J, Lontos K, Boyiadzis M. Phase 2 study of epigenetic priming with decitabine followed by cytarabine for acute myeloid leukemia in older patients. Am J Hematol. 2024 Mar;99(3):380-386. doi: 10.1002/ajh.27212. Epub 2024 Jan 22. PMID 38258329

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine + Cytarabine: Participants received decitabine 20mg/m^2 intravenously (IV) for five days followed by cytarabine 100mg/m^2 continuous IV infusion over 24 hours for five days.
Period: Overall Study
Arm/Group | Decitabine + Cytarabine
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of participants with each of the observed demographic and clinical characteristics.
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 76.2 [67.1 to 87.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0
Acute myeloid leukemia (AML) Type [Number; unit: participants]
  AML with MDS Changes | 24
  Primary AML | 12
  Treatment-Related AML | 8
Baseline ECOG Status [Number; unit: participants] — ECOG Scale (patient's level of functioning) ;0-Fully active, able to carry on all pre-disease performance without restriction;1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work;2-Ambulatory and capable of all selfcare but unable to carry out any work; activities. Up and about more than 50% of waking hours;3-Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours;4-Completely disabled. Cannot do any self-care. Totally confined to bed or chair; 5-death
  participants
    ECOG Status 0 | 7
    ECOG Status 1 | 24
    ECOG Status 2 | 13
Charlson comorbidity index [Number; unit: participants] — Charlson comorbidity index predicts the one-year mortality for a patient who may have a range of comorbid conditions. Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one. A score of >6 indicates metastatic disease/greater risk of death.
  participants
    4 | 1
    5 | 5
    6 | 20
    >6 | 18
FLT (FMS-like tyrosine kinase 3) and NPM1 (nucleophosmin) gene Status [Number; unit: participants] — European LeukemiaNet (ELN) recommendations/classifications for diagnosis and management of acute myeloid leukemia (AML) - genetic mutational (+/-) status of NPM1, FLT3-ITD genes and D835 codon.
  participants
    Favorable | 3
    Intermediate-1 | 16
    Intermediate-2 | 3
    Adverse | 22
FLT and NPM1 Status [Number; unit: participants] — FLT3 and NPM1 status was checked on 1 'Favorable', 8 'Intermediate-1' and 3 'Intermediate-2' patients
  participants
    FLT3 D835+ | 2
    FLT3-/NPM1- | 3
    FLT3-/NPM1+ | 2
    FLT3+/NPM1- | 2
    FLT3-+/NPM1+ | 2
    No data for FLT3 and NPM1 status | 33
Albumin [Median (Full Range); unit: g/dL] | 3.4 [2.0 to 4.6]
Bilirubin [Median (Full Range); unit: mg/dL] | 0.8 [0.3 to 11.8]
Creatinine [Median (Full Range); unit: mg/dL] | 0.97 [0.4 to 3.5]
Hematocrit (volume of red blood cells / total volume of blood) [Median (Full Range); unit: percentage of total blood volume] | 27.9 [17.4 to 38.9]
Lactate dehydrogenase (LDH) [Median (Full Range); unit: IU/L] | 233 [99 to 3314]
White Blood Cells (WBC) [Median (Full Range); unit: 10^9 white blood cells per liter] | 5.25 [1 to 104]
Bone marrow blasts (number of blasts/total cells in bone marrow) [Median (Full Range); unit: percent of total white blood cell count] | 56.65 [20.0 to 94.3]
Peripheral Blood blasts (number of blasts/total white blood cell count) [Median (Full Range); unit: percent] | 13 [0 to 91]
Platelets [Median (Full Range); unit: 10^9 cells per liter] | 54.5 [14 to 375]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Best Clinical Response Experienced
Description: The number of participants who experienced either a Complete Response, Complete Response with Incomplete Count Recovery, Partial Response, or Progressive Disease. Complete response: Less than 5% blasts in an aspirate sample of a patient who has an absolute neutrophil count of >1000µ/L and platelets >100,000µ/L; Complete response with incomplete count recovery: Complete response except for residual neutropenia (<1000µ/L) or thrombocytopenia (<100,000µ/L) Partial response: Decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow aspirate; Progressive disease: Failure to achieve complete response or partial response
Time Frame: Up to 38 months
Population: Evaluable participants with known Clinical Response.
Measure: Number; unit: Participants
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 39
Participants
  Complete Response | 20
  Complete Response with Incomplete Count Recovery | 6
  Partial Response | 6
  Progressive Disease | 7

2. Primary Outcome: Proportion of Participants With Clinical Response (CR)
Description: The number of participants (out of 39) who experienced Clinical Response as Complete Response, or, Complete Response + Complete Response with Incomplete Count Recovery (exact Clopper-Pearson confidence interval).
Time Frame: Up to 38 months
Population: Evaluable participants with known Clinical Response (CR) (Complete Response, Complete Response with Incomplete Count Recovery, or Partial Response), and participants who had Progressive Disease.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 39
Proportion of participants
  Complete | 0.51 [0.37 to 0.65]
  Complete + Complete with Incomplete Count Recovery | 0.67 [0.52 to 0.79]

3. Secondary Outcome: Numbers of Patients (Out of 44) Experiencing Adverse Events With CTCAE Grade ≥ 3 or Adverse Events Grade ≥ 4
Description: The number of participants (out of 44) experiencing adverse events, with CTCAE Grade ≥ 3 or Adverse Events Grade ≥ 4
Time Frame: Up to 38 months
Population: All study participants.
Measure: Number; unit: Participants
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 44
Participants
  Adverse Events Grade ≥ 3 | 44
  Adverse Events Grade ≥ 4 | 41

4. Secondary Outcome: Proportion of Participants With Survival to Four and Eight Weeks and One Year
Description: The proportion of all participants experiencing four and eight-week mortality, or, who were alive at one year.
Time Frame: Up to one year (4 weeks, 8 weeks, and one year)
Population: All study participants.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 44
Proportion of participants
  Death Within 4 Weeks | 0.023 [0.0012 to 0.10]
  Death Within 8 Weeks | 0.091 [0.032 to 0.20]
  Alive at One Year | 0.48 [0.35 to 0.61]

5. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 38 months (median follow-up = 25.4 months)
Population: All study participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 44
months | 10.8 [9.6 to 16.0]

6. Secondary Outcome: Overall Survival (OS) in Participants Who Experienced Complete Response
Time Frame: Up to 38 months (median follow-up = 25.4 months)
Population: Evaluable participants who experienced a Clinical Response (CR) of Complete Response.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 20
months | 18.9 [13.6 to NA] — Upper bound of CI not reached.

7. Secondary Outcome: Overall Survival (OS) in Participants Who Experienced Complete Response or Complete Response With Incomplete Count Recovery
Time Frame: Up to 38 months (median follow-up = 25.4 months)
Population: Evaluable participants who experienced a Clinical Response (CR) of Complete Response, or Complete Response with Incomplete Count Recovery.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 26
months | 15.7 [12.4 to 29.0]

8. Secondary Outcome: Overall Survival (OS) in Participants Who Experienced Complete Response, Complete Response With Incomplete Count Recovery, or Partial Response
Time Frame: Up to 38 months (median follow-up = 25.4 months)
Population: Evaluable participants who experienced a Clinical Response (CR) of Complete Response, Complete Response with Incomplete Count Recovery, or, Partial Response.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 32
months | 15.7 [10.6 to 21.5]

9. Secondary Outcome: Demographic Characteristics and Clinical Measures as Potential Predictors of Overall Survival (OS)
Description: Median number of months of survival per individual demographic characteristics and clinical measures.
Time Frame: Up to 38 months (median follow-up = 25.4 months)
Population: All study participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 44
months
  Age ≤ 75 years | 12.4 [10.4 to NA] — Upper bound of CI not reached.
  Age > 75 years | 9.7 [6.9 to 17]
  Sex - Female | 11.0 [9.6 to NA] — Upper bound of CI not reached.
  Sex - Male | 10.6 [6.5 to 18.9]
  ECOG status 0 | 16.0 [7.6 to NA] — Upper bound of CI not reached.
  ECOG status 1 | 12.6 [9.7 to 18.9]
  ECOG status 2 | 4.2 [1.9 to NA] — Upper bound of CI not reached.
  Charlson co-morbidity status ≤ 6 | 14.3 [10.4 to NA] — Upper bound of CI not reached.
  Charlson co-morbidity status > 6 | 7.4 [3.6 to NA] — Upper bound of CI not reached.
  FLT and NPM1 Status: favorable | 18.9 [6.9 to NA] — Upper bound of CI not reached.
  FLT and NPM1 Status: intermediate | 7.6 [4.2 to 17]
  FLT and NPM1 Status: adverse | 14.3 [10.6 to NA] — Upper bound of CI not reached.
  AML Type-Primary AML | 10.3 [4.2 to NA] — Upper bound of CI not reached.
  AML Type-AML with MDS changes | 11.5 [7.6 to 17]
  AML Type-Treatment-related AML | 12.4 [6.5 to NA] — Upper bound of CI not reached.
  WBC ≤ 5.25 µ/L | 14.9 [12.4 to NA] — Upper bound of CI not reached.
  WBC > 5.25 µ/L | 7.6 [3.6 to 16]
  Hematocrit ≤ 27.9% | 13.0 [6.9 to NA] — Upper bound of CI not reached.
  Hematocrit > 27.9% | 10.5 [7.6 to 21.5]
  Platelets ≤ 54.5 µ/L | 10.4 [5.5 to 16]
  Platelets > 54.5 µ/L | 15.4 [9.6 to NA] — Upper bound of CI not reached.
  Albumin ≤ 3.4 gm/dL | 10.8 [6.9 to 15.4]
  Albumin > 3.4 gm/dL | 13.6 [7.6 to NA] — Upper bound of CI not reached.
  Creatinine ≤ 0.97 mg/dL | 10.6 [9.6 to 17]
  Creatinine > 0.97 mg/dL | 14.9 [5.5 to NA] — Upper bound of CI not reached.
  Bilirubin ≤ 0.8 mg/dL | 10.4 [5.5 to NA] — Upper bound of CI not reached.
  Bilirubin > 0.8 mg/dL | 13.6 [7.6 to 21.5]
  LDH ≤ 233 IU/L | 14.4 [10.4 to NA] — Upper bound of CI not reached.
  LDH > 233 IU/L | 6.9 [4.2 to 16.7]
  Bone marrow blasts ≤ 53.65% | 14.9 [12.4 to 29.0]
  Bone marrow blasts > 53.65% | 7.6 [4.2 to 16.7]
  Peripheral blasts ≤ 13% | 14.0 [10.4 to NA] — Upper bound of CI not reached.
  Peripheral blasts > 13% | 7.6 [4.2 to NA] — Upper bound of CI not reached.

10. Secondary Outcome: Relapse-Free Survival in Participants With Complete Response or Complete Response With Incomplete Count Recovery.
Time Frame: Up to 38 months
Population: Evaluable participants who experienced a Clinical Response (CR) of Complete Response or Complete Response with Incomplete Count Recovery.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Decitabine + Cytarabine
Number analyzed (Participants) | 26
months | 11.7 [9.4 to 25.3]

11. Secondary Outcome: Relapse-Free Survival in Participants With Complete Response, Complete Response With Incomplete Count Recovery or Partial Response, and Received Maintenance Therapy
Time Frame: Up to 38 months
Population: Evaluable participants who experienced a Clinical Response (CR) of Complete Response, Complete Response with Incomplete Count Recovery, or Partial Response.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- Decitabine + Cytarabine + Maintenance Therapy: Participants received decitabine 20mg/m^2 intravenously (IV) for five days followed by cytarabine 100mg/m^2 continuous IV infusion over 24 hours for five days. Participants also received decitabine 20mg/m^2 IV daily for 5 days to be given as an outpatient (maintenance therapy) until disease progression (at least one cycle).
Arm/Group | Decitabine + Cytarabine + Maintenance Therapy
Number analyzed (Participants) | 29
months | 11.5 [9.4 to 25.3]

12. Secondary Outcome: Functional Assessment of Cancer Therapy: Health-related Quality of Life (HRQOL) Measure
Description: The FACT-Leu Health-related Quality of Life (HRQOL) Measure is a 27-item FACT-G scale plus a 17-item leukemia sub-scale. The FACT-G contains uses Likert scale 0-4, with 0 ="not at all" and 4 ="very much". The total score can be 0-108 and includes 7 items related Physical Well-being (PWB), 7 items related to Social Well-being (SWB), 6 items related to Emotional Well-being (EWB) and 7 items related to Functional Well-Being (FWB). Higher scores are better. Responses based on how patients felt in the past 7 days. FACT-Leu uses a Likert scale (0 to 4, with 0= "not at all" and 4= "very much"). The total score for the 17 items can be 0-68. Higher scores are better. The FACT-Leu total is the sum of FACT-G and FACT Leu and ranges from 0-176. Higher scores are better. FACT Trial Outcome Index is derived by adding scores on the PWB and FWB sub-scales to the leukemia sub-scales. The total for this index score is from 0-124. Higher scores are better.
Time Frame: Baseline to Post-treatment, up to 5 years
Population: Participants that received at least one cycle of treatment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Decitabine + Cytarabine + Maintenance Therapy
Number analyzed (Participants) | 35
units on a scale
  Baseline FACT-LEU Subscale | 52.05 (1.68)
  Baseline FACT Trial Outcome Index | 92.90 (3.60)
  Baseline FACT-LEU Total | 135.40 (3.90)
  Baseline FACT-G Total | 83.57 (2.44)
  Baseline FACT-G - Physical Well-Being | 22.75 (1.12)
  Baseline FACT-G - Social Well-Being | 24.73 (0.66)
  Baseline FACT-G - Emotional Well-Being | 17.30 (0.77)
  Baseline FACT-G - Functional Well-Being | 17.16 (1.26)
  Post-treatment LEU Subscale | 51.78 (1.39)
  Post-treatment FACT Trial Outcome Index | 92.50 (3.21)
  Post-treatment FACT-LEU Total | 137.26 (3.97)
  Post-treatment FACT-G Total | 84.23 (2.73)
  Post-treatment FACT-G - Physical Well-Being | 23.20 (0.75)
  Post-treatment FACT-G - Social Well-Being | 24.72 (0.74)
  Post-treatment FACT-G - Emotional Well-Being | 18.07 (0.86)
  Post-treatment FACT-G - Functional Well-Being | 16.62 (1.46)

ADVERSE EVENTS:
Arm/Group | Decitabine + Cytarabine
Serious Adverse Events (participants affected / at risk) | 30/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine + Cytarabine (N=44)
Anemia (Blood and lymphatic system disorders) | 3
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Chest pain - cardiac (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 2
Fever (General disorders) | 2
General disorders and administration site conditions (General disorders) | 1
Malaise (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 1
Infections and infestations (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1
Creatinine increased (Investigations) | 2
INR increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal and urinary disorders (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine + Cytarabine (N=44)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 32
Febrile neutropenia (Blood and lymphatic system disorders) | 34
Atrial fibrillation (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 3
Pericardial effusion (Cardiac disorders) | 4
Sinus tachycardia (Cardiac disorders) | 4
Eye disorders (Eye disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 3
Gastrointestinal disorders (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 18
General disorders and administration site conditions (General disorders) | 6
Non-cardiac chest pain (General disorders) | 6
Pain (General disorders) | 8
Chills (General disorders) | 10
Fever (General disorders) | 11
Fatigue (General disorders) | 19
Edema limbs (General disorders) | 21
Bronchial infection (Infections and infestations) | 3
Enterocolitis infectious (Infections and infestations) | 3
Mucosal infection (Infections and infestations) | 4
Skin infection (Infections and infestations) | 4
Infections and infestations (Infections and infestations) | 8
Lung infection (Infections and infestations) | 17
Investigations (Investigations) | 5
Creatinine increased (Investigations) | 8
Activated partial thromboplastin time prolonged (Investigations) | 10
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 10
Alanine aminotransferase increased (Investigations) | 11
INR increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 14
Lymphocyte count decreased (Investigations) | 23
Neutrophil count decreased (Investigations) | 25
White blood cell decreased (Investigations) | 34
Platelet count decreased (Investigations) | 35
Anorexia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 16
Hypokalemia (Metabolism and nutrition disorders) | 23
Hyponatremia (Metabolism and nutrition disorders) | 25
Hypoalbuminemia (Metabolism and nutrition disorders) | 27
Back pain (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 10
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 5
Hematuria (Renal and urinary disorders) | 14
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15
Alopecia (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 7
Hematoma (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3
Vascular disorders (Vascular disorders) | 4
Hypertension (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes